CLINICAL TRIAL: NCT03360825
Title: Electrophysiological Comparison of mAP and mADM Using EMG
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Assistant Professor of Anesthesiology, College of Medicine, Mayo Clinic
Other Study IDs: 17-006680
Record Dates: First submitted 2017-11-22; First posted 2017-12-04 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TetraGraph — The TetraGraph is a dedicated neuromuscular stimulator / recorder intended to evoke, record, and analyze muscle action potentials during surgical procedures

SUMMARY:
The primary aim of this clinical investigation is to examine a prototype of a quantitative monitoring instrument that will meet most, if not all, of the clinical requirements.

DETAILED DESCRIPTION:
This is a blinded, single-center, prospective study in patients during surgery, requiring use of neuromuscular blockade. Neurostimulation will be used to monitor objective responses, as per current clinical routine. Data collection of Tetragraph EMG responses will be unavailable to the clinician for clinical decision-making, as per current clinical routine, but will be stored on the interfaced SD card.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older.
2. American Society of Anesthesiology (ASA) physical status I-III criteria (Table I).
3. Subject has provided verbal consent
4. BMI <39

Exclusion Criteria

1. Presence of an underlying neuromuscular disease.
2. Presence of renal or hepatic disease.
3. Subject has open skin sores in the locations needed for electrode application (forearms).
4. Patients on oral anticholinesterase, anti-seizure medications, and magnesium sulfate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for this study includes patients receiving neuromuscular blocking agents during a surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Primary performance assessment of TetraGraph device | Duration of surgery
  Agreement between the mAP and mADM EMG based TOF ratios
Primary performance assessment of TetraGraph device | Duration of surgery
  Agreement between the mAP and mADM EMG based TOF counts

SECONDARY OUTCOMES:
Secondary performance assessment of TetraGraph device | Duration of surgery
  Correlation between stimulation current and T1 twitch height in the two muscles
Secondary performance assessment of TetraGraph device | Duration of surgery
  Comparison of EMG to the quantitative AMG monitor

CONTACTS AND LOCATIONS:
Overall Officials: J R Renew, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gatke MR, Viby-Mogensen J, Rosenstock C, Jensen FS, Skovgaard LT. Postoperative muscle paralysis after rocuronium: less residual block when acceleromyography is used. Acta Anaesthesiol Scand. 2002 Feb;46(2):207-13. doi: 10.1034/j.1399-6576.2002.460216.x. PMID 11942873
- [Background] Cammu G, De Witte J, De Veylder J, Byttebier G, Vandeput D, Foubert L, Vandenbroucke G, Deloof T. Postoperative residual paralysis in outpatients versus inpatients. Anesth Analg. 2006 Feb;102(2):426-9. doi: 10.1213/01.ane.0000195543.61123.1f. PMID 16428537
- [Background] Kim KS, Lew SH, Cho HY, Cheong MA. Residual paralysis induced by either vecuronium or rocuronium after reversal with pyridostigmine. Anesth Analg. 2002 Dec;95(6):1656-60, table of contents. doi: 10.1097/00000539-200212000-00033. PMID 12456433
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Nisman M. Intraoperative acceleromyographic monitoring reduces the risk of residual neuromuscular blockade and adverse respiratory events in the postanesthesia care unit. Anesthesiology. 2008 Sep;109(3):389-98. doi: 10.1097/ALN.0b013e318182af3b. PMID 18719436
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Vender JS, Gray J, Landry E, Gupta DK. Intraoperative acceleromyography monitoring reduces symptoms of muscle weakness and improves quality of recovery in the early postoperative period. Anesthesiology. 2011 Nov;115(5):946-54. doi: 10.1097/ALN.0b013e3182342840. PMID 21946094
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Hemmerling TM, Le N. Brief review: Neuromuscular monitoring: an update for the clinician. Can J Anaesth. 2007 Jan;54(1):58-72. doi: 10.1007/BF03021901. PMID 17197470
- [Background] Brull SJ, Silverman DG. Visual and tactile assessment of neuromuscular fade. Anesth Analg. 1993 Aug;77(2):352-5. doi: 10.1213/00000539-199308000-00024. PMID 8394051
- [Background] Grayling M, Sweeney BP. Recovery from neuromuscular blockade: a survey of practice. Anaesthesia. 2007 Aug;62(8):806-9. doi: 10.1111/j.1365-2044.2007.05101.x. PMID 17635429
- [Background] Claudius C, Viby-Mogensen J. Acceleromyography for use in scientific and clinical practice: a systematic review of the evidence. Anesthesiology. 2008 Jun;108(6):1117-40. doi: 10.1097/ALN.0b013e318173f62f. PMID 18497614
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Connelly NR, Silverman DG, O'Connor TZ, Brull SJ. Subjective responses to train-of-four and double burst stimulation in awake patients. Anesth Analg. 1990 Jun;70(6):650-3. doi: 10.1213/00000539-199006000-00012. PMID 2160781
- [Background] CHURCHILL-DAVIDSON HC, RICHARDSON AT. The action of decamethonium iodide (C.10) in myasthenia gravis. J Neurol Neurosurg Psychiatry. 1952 May;15(2):129-33. doi: 10.1136/jnnp.15.2.129. No abstract available. PMID 14928082
- [Background] Liang SS, Stewart PA, Phillips S. An ipsilateral comparison of acceleromyography and electromyography during recovery from nondepolarizing neuromuscular block under general anesthesia in humans. Anesth Analg. 2013 Aug;117(2):373-9. doi: 10.1213/ANE.0b013e3182937fc4. Epub 2013 Jul 2. PMID 23821356
- [Background] Phillips S, Stewart PA, Freelander N, Heller G. Comparison of evoked electromyography in three muscles of the hand during recovery from non-depolarising neuromuscular blockade. Anaesth Intensive Care. 2012 Jul;40(4):690-6. doi: 10.1177/0310057X1204000416. PMID 22813498